CLINICAL TRIAL: NCT02283112
Title: Validation of Drug Assays in Various Biological Matrices
Status: Recruiting | Type: Observational
Sponsor: Helen Reynolds (Other)
Responsible Party: Sponsor-Investigator, Helen Reynolds, Research nurse, University of Liverpool
Organization: University of Liverpool (Other)
Other Study IDs: RLUH 4520
Record Dates: First submitted 2014-10-29; First posted 2014-11-05 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Antiviral Agents; Anti-Infective Agents; Contraceptives, Oral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: antivirals, antimicrobials, oral contraceptive, erectile dysfunction agents

SUMMARY:
This study aims to ensure that assays that measure drug concentrations are accurate and precise in different matrices when quantified using high performance liquid chromatography -tandem mass spectrometry (HPLC-MS/MS). The study involves collecting samples of various bodily fluids to quantify antimicrobials, antivirals, oral contraceptives and erectile dysfunction agents. Samples will also be obtained from individuals not receiving these medications for quality control purposes.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age

Exclusion Criteria:

* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers receiving specific medication or healthy volunteers taking no medication.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To measure drug concentrations using high performance liquid chromatography -tandem mass spectrometry (HPLC-MS/MS) (accuracy and precision of assays that measure drug concentrations) | Follow up up to 5 years
  Assay validation

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Liverpool & Broadgreen Univeristy Hospitals NHS Trust, Liverpool, United Kingdom